CLINICAL TRIAL: NCT06211023
Title: An Open-label, Randomized, Controlled, Phase II/III Study of SHR-A1921 With or Without Carboplatin Verus Investigator's Choice of Platinum-based Doublet Chemotherapy in Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: A Study of SHR-A1921 With or Without Carboplatin in Subjects With Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-301
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Intervention Model Description: SHR-A1921 with or without Carboplatin compared with Investigator's Choice of Platinum-based Doublet Chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1: SHR-1921 (Experimental)
  Interventions: Drug: SHR-1921
- Treatment group 2: SHR-1921 + carboplatin dose level 1 (Experimental)
  Interventions: Drug: carboplatin
- Treatment group 3: SHR-1921 + carboplatin dose level 2 (Experimental)
  Interventions: Drug: carboplatin
- Treatment group 4: platinum-based doublet chemotherapy (Other)
  Interventions: Drug: platinum-based doublet chemotherapy

INTERVENTIONS:
Drug: SHR-1921 — SHR-1921
  Arms: Treatment group 1: SHR-1921
Drug: carboplatin — carboplatin AUC 4
  Arms: Treatment group 2: SHR-1921 + carboplatin dose level 1
Drug: carboplatin — carboplatin AUC 5
  Arms: Treatment group 3: SHR-1921 + carboplatin dose level 2
Drug: platinum-based doublet chemotherapy — platinum-based doublet chemotherapy
  Arms: Treatment group 4: platinum-based doublet chemotherapy

SUMMARY:
This is an open-label, randomized, controlled, two-part study to evaluate the safety and efficacy of SHR-A1921 with or without carboplatin verus investigator's choice of platinum-based doublet chemotherapy in subjects with recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. Be able to provide fresh or archived tumour tissue.
3. Pathologically diagnosed epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
4. At least one measurable lesion according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
6. With a life expectancy ≥ 12 weeks.
7. Adequate bone marrow reserve and organ function.

Exclusion Criteria:

1. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion with clinical symptoms.
2. Previous or co-existing malignancies.
3. Has a history of non-infectious ILD/pneumonitis that required steroids, or has current ILD/pneumonitis;
4. Subjects with active hepatitis B or active hepatitis C;
5. Subjects who have received systemic anti-tumor treatments 4 weeks prior to the initiation of the study treatment.
6. Subjects who have been treated with TOP1 inhibitors, TROP-2 ADC or ADCs with TOP1 inhibitors as payload.
7. Has unresolved CTCAE ≥grade 2 toxicities from previous anticancer therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate Assessed by Investigator According to RECIST v1.1 | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Duration of Response (DoR) Assessed by Investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Disease Control Rate (DCR) Assessed by Investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Progression-Free Survival (PFS) Assessed by Investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Overall Survival (OS) | Screening up to study completion, an average of 1 year
CA-125 Response assessed by the Gynecologic Cancer Intergroup (GCIG) criteria | Screening up to study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided